CLINICAL TRIAL: NCT02096809
Title: Evaluation of Soft Tissue Healing and Implant Stability of Cochlear Baha BI300/BA400 Implant System Loaded From 1 Week Post-surgery After Linear Incision Without Soft Tissue Reduction.
Brief Title: Stability of the Cochlear Baha BI300/BA400 Implant System Loaded From 1 Week Post-surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Lars Vendelbo Johansen, Consultant, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-5-14; 1-10-72-5-14 (Other: Central DK Region Committees on Health Research Ethics)
Record Dates: First submitted 2014-03-23; First posted 2014-03-26 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Hearing Loss - Conductive
Keywords: Bone Conduction; Hearing loss - conductive; Osseointegration; Prostheses and Implants
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One week loading of Bone Anchored Hearing Aid (BAHA) (Experimental): Bone Anchored Hearing Aid (BAHA) loading after one week
  Interventions: Procedure: One week loading of Bone Anchored Hearing Aid (BAHA); Device: Cochlear Baha BI300/BA400 Implant System

INTERVENTIONS:
Procedure: One week loading of Bone Anchored Hearing Aid (BAHA) — Patients in this arm will be fitted with the BAHA one week after surgery.
Device: Cochlear Baha BI300/BA400 Implant System

SUMMARY:
Objectives

* To evaluate the safety of processor loading of the Cochlear BI300/BA400 implant system 1 week after implantation
* To evaluate the short term soft tissue healing and the long term skin reaction, with the new Cochlear BI300/BA400 implant system using the linear incision without subcutaneous tissue reduction.
* To produce reference data regarding the stability of the BI300/BA400 implant system.

Study design: Prospective cohort study. Patients: 24 adults with anticipated normal skin and bone quality eligible for bone anchored implant surgery.

Intervention: Loading of the sound processor one week after surgery Main outcome measures: Implant stability, soft tissue reaction, skin overgrowth, pain and numbness will be assessed.

It is hypothesized that implant loading can be performed one week after surgery without any changes in implant stability, soft tissue reaction, skin overgrowth, pain or numbness around implant.

DETAILED DESCRIPTION:
Background Implant stability

Until recently, the implants used in Baha surgery have exclusively been standard Brånemark type of titanium implants with an as-machined surface finish. The recommended procedure for Baha implantation with the machined titanium implants uses a 12-week healing period before loading the implant with a sound processor, in order to allow sufficient time for the implant to become integrated in the bone. The Cochlear Baha BI300 Series implant was designed to improve implant stability at placement and over time, thus making it possible to reduce the time to sound processor fitting. The implant features a wider diameter compared to the previous generation Baha implant, small-sized threads at the cylindrical portion of the implant underneath the flange, and a roughened implant surface due to formation of titanium oxide after blasting.

Six-month data from a multi-centre clinical investigation comparing the new implant with the previous generation Baha implant using a 6-week loading protocol, shows significantly higher Implant Stability Quotient (ISQ) values (measured by resonance frequency analysis) for the new implant at each time point, and no reduction in stability after loading (Dun et al., 2011). The data from the study suggest that the implant stability achieved 6 weeks after implantation is sufficient to support the sound processor. The data also suggest that a further reduction of the time to sound processor fitting may be possible, provided favourable bone conditions at the implant site and provided satisfactory soft tissue status at the time of loading. Hence, a clinical investigation with implant loading 21 days post-surgery was initiated by the team in Nijmegen, and 6-month data from the investigation confirm that it is safe to attach the sound processor after 3 weeks (Faber et al., 2012). Early results from two other studies using loading times of 4 weeks (McLarnon et al., 2012) and 2 weeks (Green et al., 2011), respectively, have also been presented and show good outcomes. All studies have been performed on patients with good bone quality.

Data from a prospective study with 49 patients loaded from 2 weeks post-surgery show no initial dip in stability and show no decrease in stability in the period after processor loading (ongoing study, awaiting publication). The stability of the implant in this study after one week is sufficient for processor loading at this time. No studies exist that investigates the effect on stability after processor loading 1 week postoperatively.

Implant stability measurement

The method of choice for implant stability measurements uses resonance frequency analysis (RFA) of a small magnetic rod attached to the abutment at the time of measuring (Osstell A/B, Gothenburg, Sweden). However, this method returns a number (Implant Stability Quotient, ISQ) for the stability that is dependent on the length of the abutment attached to the implant. To our knowledge there exists no clinical data that correlates the stability measurements made with different abutment length.

Soft tissue management

For three decades, the recommended procedure for Baha implantation advocated a hair free transplant measuring 25 x 25 mm placed direct on the periosteum. The purpose is to obtain an immobile skin, hence reducing the risk of adverse skin reactions in the area. Since there is no or only weak adherence between the abutment and surrounding soft tissue it is anticipated that, if no skin reduction is performed, epidermal down growth and pocket formation may occur over time, increasing the risk for infection in the implant area. This surgical procedure, with skin transplant, has proven safe; however, skin complications still occur and account for the majority of reported complications with Baha implants.

The newly introduced Cochlear BA400 abutment is covered with hydroxyapatite at the area of the abutment touching the skin and subcutaneous tissues. The abutment has been approved for surgery using a less invasive surgical technique (linear incision without subcutaneous tissue reduction) (www.cochlear.com). It has been shown in animal studies that the hydroxyapatite coating favours soft tissue healing without pocket formation (Larsson et al, 2012).

To our knowledge there exists no studies that compare the results with the BA400 inserted using the linear incision without subcutaneous tissue reduction with other abutments using the same technique.

Objectives

* To evaluate the safety of processor loading of the Cochlear BI300/BA400 implant system 1 week after implantation
* To evaluate the short term soft tissue healing and the long term skin reaction, with the new Cochlear BI300/BA400 implant system using the linear incision without subcutaneous tissue reduction.
* To produce reference data regarding the stability of the BI300/BA400 implant system.

IMPLANT DEVICE

The following Conformité Européenne (CE) marked implant with pre-mounted abutment will be used (MDD Class IIb medical devices, manufacturer: Cochlear Bone Anchored Solutions, Mölnlycke, Sweden):

• Cochlear Baha BI300 4 mm with Cochlear BA400 Abutment (DermalockTM). Length of the abutment will be decided after measuring the thickness of the skin with a specific tool.

TREATMENT

Surgery The implants will be placed according to the procedure for one-stage surgery. The surgical procedure is by a linear incision without removal of subcutaneous tissue. The implant will be places outside the linear incision. Only in cases where the longest available abutment (12mm) is deemed too short there will be performed a minimal soft tissue reduction of subcutaneous fatty tissue. A 5 mm punch will be used to punch the hole for the abutment in the skin flap.

All patients will receive treatment, thus no placebo control group is used. The surgical technique is the one recommended by the manufacturer for this type of implant and hence the study does not introduce any new surgical techniques or modifications hereof.

The risks with this treatment are: bleeding per- and postoperatively, wound infection and damage to surrounding tissues including sensory nerves to the scalp and loss of the implant. These risks are well known risks with known treatments and the study introduces no new risks.

Sound processor loading Sound processor fitting and loading will be performed 1 week after implant surgery, or at the discretion of the investigator. The decision to load an implant will be based on assessment of implant stability and status of the soft tissue. Patients who are evaluated as not ready to be loaded 1 week after surgery will be loaded as soon as the healing is sufficient.

ETHICAL CONSIDERATIONS There are no known extra risks or adverse effects of the new abutment compared to the previous abutment supplied by the manufacturer of the implant. Preliminary results (7) have shown promising positive effects on the soft tissue healing and implant stability. In conclusion, the new abutment design have the same potential adverse effects. All patients are offered the new abutment system.

The surgical technique: linear incision without soft tissue reduction, is recommended by the manufacturer to use with this implant system.

Stability measurements with radio frequency analysis have no known side effects.

The stability of the implant at the planned loading time (1 week) has been shown in previous studies to be better than that at which earlier generation implants has been loaded after 6 weeks(Dun et al., 2011,8). However, loading of the implant 1 week post-surgery has the potential risk of influencing the osseous integration of the implant in the cranial bone which could lead to loosening of the implant and eventually loss of implant. The patients will be controlled with stability measurement 1 week after loading of the implant and a possible loosening of the implant can be taken care of.

Loading of the implant 1 week post-surgery has potential benefits for the patient in the form of faster audiological rehabilitation and fewer visits to the hospital.

No specific recruitment of patients is made in this study. Patients referred to the hospital for Baha-surgery are evaluated according to the inclusion criteria and all patients (within the inclusion period) that are included are offered to be part of the study group.

Patients will be invited with a letter to a clinical examination prior to the operation. In this letter all patients are requested to bring an assessor if deemed necessary.

If the patient meets the inclusion criteria, spoken and written information about the study will be given by one of the investigators at the out-patient clinic. The examination and information will take place in a state-of-the-art examination room with no interruptions and there will be given time to discuss all relevant details of the study and questions will be answered.

The informed consent should be signed before the day of surgery. There will be approximately three weeks between the written information and the expected informed consent and questions can be answered in this period by contacting the investigators by e-mail or phone. If the patient decides not to participate in the study he will still be offered the operation with the same procedure, but the loading time will follow standard recommendations and no extra stability measurements will be performed.

SAMPLE SIZE CALCULATION To detect a difference in ISQ between baseline and any measurement point during follow up of 4 ISQ points, the study needs 21 patients in each group, not accounting for drop-out (comparison of two means, st.d.=4 in each group (5), α=0,05 two-sided, power=90%). To allow for a drop-out rate of around 10%, we include 25 patients. The time estimated to include this number of patients is 3 months.

With 25 patients we will be able to detect a risk difference of 0,41 for having Holgers' index 0 or 1-4 in the two groups (comparison of two proportions, α=0,05 two-sided, power=90%).

STATISTICS

Results will be analysed on the basis of both descriptive and inferential statistics.

The following results will be reported

* Baseline characteristics
* Implant stability by visit, represented as a Line plot of Mean ISQ (95% confidence interval).
* Difference of the mean ISQ between intervention and control group at each measurement point (students t-test).
* Average implant stability, as assessed by the mean area under the curve of ISQ-measurements (mean, confidence interval).
* Effect of implant loading on implant stability, as assessed by change in Mean ISQ from time of loading to subsequent visit(s) (paired t-tests, confidence interval).
* Soft tissue reactions (Holgers' Index) at each measurement point (Mantel-Haenszel statistics)
* Soft tissue overgrowth at each measurement point (Mantel-Haenszel statistics)
* Presence of pain at each measurement point (Mantel-Haenszel statistics).
* Presence of numbness at each measurement point (Mantel-Haenszel statistics).
* Dichotomization of the Holgers' scale will be performed by categorizing Holgers' grade 0 and 1 as "No clinically significant tissue reaction" and Holgers' grade 2-5 as "Clinically significant tissue reaction" and comparisons made between groups with the Fischer exact test.
* Implant loss, as assessed by survival analysis (if any).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age, with normal intelligence.
* Absence of previous radiotherapy to the implant area.
* Absence of active skin disease in the implant area.
* Absence of diabetes.
* Absence of osteoporosis
* Absence of any relevant medical history or current disease/treatment/medication that may affect bone or skin quality in the implant area.

Exclusion Criteria:

* No further

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Implant stability | Day of surgery
  Implant stability quotient measured at day of surgery. Implant stability is assessed using resonance frequency analysis. The measurement renders Implant Stability Quotient (ISQ) values from 1 to 100. Two perpendicular measurements are performed at each implant. The highest and lowest ISQ value out of three measurements obtained at each time point will be recorded. Measurements will be performed at the abutment level, and the Osstell ISQ instrument and SmartPeg Type 55 (Osstell, Gothenburg, Sweden) will be used.
Implant stability | One week
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.
Implant stability | Two weeks
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.
Implant stability | One month
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.
Implant stability | 3 months
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.
Implant stability | 6 months
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.
Implant stability | 12 months
  See description for Implant stability, day of surgery Implant stability is assessed using resonance frequency analysis.

SECONDARY OUTCOMES:
Soft tissue status | One week
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Soft tissue status | Two weeks
  See description for soft tissue status, one week.
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Soft tissue status | One month
  See description for soft tissue status, one week.
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Soft tissue status | 3 months
  See description for soft tissue status, one week.
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Soft tissue status | 6 months
  See description for soft tissue status, one week.
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Soft tissue status | 12 months
  See description for soft tissue status, one week.
  0. No irritation: epithelial debris removed if present.
  1. Slight redness: temporary local treatment indicated.
  2. Red and slightly moist; no granulation tissue present.
  3. Red and moist with granulation tissue, skin overgrowth, or scar formation: Local treatment indicated.
  4. Extensive granulation, skin overgrowth, or scar formation requiring revision surgery.
  5. Removal of skin-penetrating abutment necessary to control infection.
Skin overgrowth | One week
  0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Skin overgrowth | Two weeks
  See description for skin overgrowth, one week. 0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Skin overgrowth | One month
  See description for skin overgrowth, one week. 0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Skin overgrowth | 3 months
  See description for skin overgrowth, one week. 0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Skin overgrowth | 6 months
  See description for skin overgrowth, one week. 0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Skin overgrowth | 12 months
  See description for skin overgrowth, one week. 0. No soft tissue thickening or overgrowth,
  1. Slight soft tissue thickening or overgrowth,
  2. Moderate soft tissue thickening or overgrowth. Local treatment and extra controls as indicated,
  3. Marked/distinct soft tissue thickening or overgrowth. Revision surgery is indicated.
Pain around implant | One week
  Pain will be assessed using categories based on a VAS from 0-10:
  * None 0
  * Mild 1-3
  * Moderate 4-6
  * Extensive 7-10
Pain around implant | Two weeks
  See description for pain around implant, one week
  None 0 Mild 1-3 Moderate 4-6 Extensive 7-10
Pain around implant | One month
  See description for pain around implant, one week
  None 0 Mild 1-3 Moderate 4-6 Extensive 7-10
Pain around implant | 3 months
  See description for pain around implant, one week
  None 0 Mild 1-3 Moderate 4-6 Extensive 7-10
Pain around implant | 6 months
  See description for pain around implant, one week
  None 0 Mild 1-3 Moderate 4-6 Extensive 7-10
Pain around implant | 12 months
  See description for pain around implant, one week
  None 0 Mild 1-3 Moderate 4-6 Extensive 7-10
Numbness around implant | One week
  Numbness will be assessed using categories based on a measurement of the largest distance from the abutment with altered or no sensitivity:
  * None ≤ 1cm
  * Mild 1 - 3cm
  * Moderate 3 - 5 cm
  * Extensive ≥ 5cm
Numbness around implant | Two weeks
  See description fot numbness around implant, one week
  None ≤ 1cm Mild 1 - 3cm Moderate 3 - 5 cm Extensive ≥ 5cm
Numbness around implant | One month
  See description fot numbness around implant, one week
  None ≤ 1cm Mild 1 - 3cm Moderate 3 - 5 cm Extensive ≥ 5cm
Numbness around implant | 3 months
  See description fot numbness around implant, one week
  None ≤ 1cm Mild 1 - 3cm Moderate 3 - 5 cm Extensive ≥ 5cm
Numbness around implant | 6 months
  See description fot numbness around implant, one week
  None ≤ 1cm Mild 1 - 3cm Moderate 3 - 5 cm Extensive ≥ 5cm
Numbness around implant | 12 months
  See description fot numbness around implant, one week
  None ≤ 1cm Mild 1 - 3cm Moderate 3 - 5 cm Extensive ≥ 5cm

OTHER OUTCOMES:
Implant loss | Up to one year
  Number of implants lost during the first year of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Johansen, D.MSc., Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, ENT-department, Aarhus, Denmark

REFERENCES:
- [Background] Dun CA, de Wolf MJ, Hol MK, Wigren S, Eeg-Olofsson M, Green K, Karlsmo A, Flynn MC, Stalfors J, Rothera M, Mylanus EA, Cremers CW. Stability, survival, and tolerability of a novel baha implant system: six-month data from a multicenter clinical investigation. Otol Neurotol. 2011 Aug;32(6):1001-7. doi: 10.1097/MAO.0b013e3182267e9c. PMID 21725257
- [Background] Larsson A, Wigren S, Andersson M, Ekeroth G, Flynn M, Nannmark U. Histologic evaluation of soft tissue integration of experimental abutments for bone anchored hearing implants using surgery without soft tissue reduction. Otol Neurotol. 2012 Oct;33(8):1445-51. doi: 10.1097/MAO.0b013e318268d4e0. PMID 22918110
- [Background] Faber HT, Dun CA, Nelissen RC, Mylanus EA, Cremers CW, Hol MK. Bone-anchored hearing implant loading at 3 weeks: stability and tolerability after 6 months. Otol Neurotol. 2013 Jan;34(1):104-10. doi: 10.1097/MAO.0b013e318277a282. PMID 23202148
- [Background] Holgers KM, Tjellstrom A, Bjursten LM, Erlandsson BE. Soft tissue reactions around percutaneous implants: a clinical study of soft tissue conditions around skin-penetrating titanium implants for bone-anchored hearing aids. Am J Otol. 1988 Jan;9(1):56-9. PMID 3364537
- [Background] Wazen JJ, Young DL, Farrugia MC, Chandrasekhar SS, Ghossaini SN, Borik J, Soneru C, Spitzer JB. Successes and complications of the Baha system. Otol Neurotol. 2008 Dec;29(8):1115-9. doi: 10.1097/MAO.0b013e318187e186. PMID 18833013
- [Background] McLarnon CM, Johnson I, Davison T, Hill J, Henderson B, Leese D, Marley S. Evidence for early loading of osseointegrated implants for bone conduction at 4 weeks. Otol Neurotol. 2012 Dec;33(9):1578-82. doi: 10.1097/MAO.0b013e31826dba5f. PMID 23069746